CLINICAL TRIAL: NCT04336254
Title: Safety and Efficacy Study of Allogeneic Human Dental Pulp Mesenchymal Stem Cells to Treat Severe Pneumonia of COVID-19：a Single-center, Prospective, Randomised Clinical Trial
Brief Title: Safety and Efficacy Study of Allogeneic Human Dental Pulp Mesenchymal Stem Cells to Treat Severe COVID-19 Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Beijing SH Bio-Tech Corporation, Beijing (CN) (Unknown); Utooth Biological Technology Co., Ltd. Hubei (CN) (Unknown)
Responsible Party: Principal Investigator, Ye Qingsong, Professor, Director, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020K-G005; hDPSC-CoVID-2019-02-2020 (Other: Renmin Hospital of Wuhan University)
Record Dates: First submitted 2020-03-28; First posted 2020-04-07 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: Cronovirus; Human Dental Pulp Stem Cells; Dental Stem Cell Banking
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hDPSCs group (Experimental): Routine treatment + Intravenous injection of human dental pulp stem cells
  Interventions: Biological: allogeneic human dental pulp stem cells (BSH BTC & Utooth BTC)
- Control group (Placebo Comparator): Routine treatment + Intravenous saline injection (Placebo)
  Interventions: Other: Intravenous saline injection (Placebo)

INTERVENTIONS:
Biological: allogeneic human dental pulp stem cells (BSH BTC & Utooth BTC) — Intravenous injection of 3.0x10e7 human dental pulp stem cells solution (30ml) on day 1, day 4 and day 7, based on routine treatment of COVID-19
  Arms: hDPSCs group
Other: Intravenous saline injection (Placebo) — Intravenous injection of 3ml of 0.9% saline on day 1, day 4 and day 7, based on routine treatment of COVID-19
  Arms: Control group

SUMMARY:
This clinical trial is set out to evaluate the safety and efficacy of allogeneic human dental pulp mesenchymal stem cells in the treatment of severe pneumonia caused by COVID-19; to explore the effects of human dental pulp mesenchymal stem cells in the treatment of severe pneumonia of COVID-19 in terms of reducing mortality and improving clinical prognosis; and to discover a new therapeutic strategy for COVID-19 using allogeneic human dental pulp mesenchymal stem cells.

DETAILED DESCRIPTION:
This clinical trial is set out to evaluate the followings:

1. the safety and efficacy of allogeneic human dental pulp mesenchymal stem cells in the treatment of severe pneumonia caused by COVID-19;
2. to explore the effects of human dental pulp mesenchymal stem cells in the treatment of severe pneumonia of COVID-19 in terms of reducing mortality and improving clinical prognosis; and
3. to discover a new therapeutic strategy for COVID-19 using allogeneic human dental pulp mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years;
2. Voluntarily participate in this clinical trial and sign off "informed consent form";
3. Diagnosed with severe pneumonia of COVID: respiratory distress, RR >30 times / min; resting oxygen saturation of 93% or less; arterial partial pressure of oxygen / oxygen concentration 300mmHg; SARS-CoV-2 nucleic acid test was positive.
4. Chest imaging confirm COVID-19 featured lesions in lung.

Exclusion Criteria:

1. Receive any clinical trial drug treatment for COVID-2019 within 30 days before the screening assessment;
2. Severe liver disease (e.g., Child Pugh score >=C or AST> 5 times of the upper limit);
3. Patients with known severe renal insufficiency (estimated glomerular filtration rate <=30mL / min/1.73 m2) or patients receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis;
4. Co-infection of HIV, hepatitis B, tuberculosis, influenza virus, adenovirus or other respiratory infection viruses;
5. Female patients who have no sexual protection in the last 30 days prior to the screening assessment;
6. Pregnant or lactating women or women using estrogen contraception;
7. Patients who are planning to become pregnant during the study period or within 6 months after the end of the study period;
8. Other conditions that the researchers consider not suitable for participating in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
TTCI | 1-28 days
  Time to Clinical Improvement

SECONDARY OUTCOMES:
Lung lesion | 1-28 days
  Lung Lesion by CT
Immune function | 1-28 days
  1. Th1 cytokines: IL-1β, IL- 2, TNF-a, ITN-γ;
  2. Th2 cytokines: IL- 4, IL- 6, IL- 10;
  3. Immunoglobulins: IgA, IgG, IgM, and total IgE;
  4. Lymphocyte counts: CD3+, CD4+, CD8+, CD16+,CD19+, CD56+.
Time of SARS-CoV-2 clearance | 1-28 days
  Time of SARS-CoV-2 test turns negative
Blood test | 1-28 days
  Blood cell count and classification
SPO2 | 1-28 days
  Pulse oximetry
RR | 1-28 days
  Respiratory rate
Body temperature | 1-28 days
  Body temperature
Side effects in the treatment group | 1-28 days
  Number of the included patients with hDPSCs-related adverse events, e.g. liver or kidney function failure
C-reactive protein (mg/L) | 1-28 days
  C-reactive protein in microgram per litre

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Qingsong Ye, PhD,DDS, Study Chair — Center for Regenerative Medicine, Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University (East Campus), Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye Q, Wang H, Xia X, Zhou C, Liu Z, Xia ZE, Zhang Z, Zhao Y, Yehenala J, Wang S, Zhou G, Hu K, Wu B, Wu CT, Wang S, He Y. Safety and efficacy assessment of allogeneic human dental pulp stem cells to treat patients with severe COVID-19: structured summary of a study protocol for a randomized controlled trial (Phase I / II). Trials. 2020 Jun 12;21(1):520. doi: 10.1186/s13063-020-04380-5. PMID 32532356